CLINICAL TRIAL: NCT04712539
Title: Efficacy of Combination Baloxovir and Oseltamivir Therapy in Influenza Infected Immunocompromised Hosts
Brief Title: Baloxavir and Oseltamivir for the Treatment of Severe Influenza Infection in Immunocompromised Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-0919; NCI-2020-13918 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0919 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-01

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Influenza
MeSH Terms: conditions — Hematologic Neoplasms; Influenza, Human | interventions — baloxavir; Oseltamivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (oseltamivir, baloxavir marboxil) (Experimental): Patients receive oseltamivir PO BID for up to 10 days and baloxavir marboxil PO every 72 hours for a total of 3 doses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Baloxavir Marboxil; Drug: Oseltamivir
- Arm II (oseltamivir) (Active Comparator): Patients receive oseltamivir PO BID for up to 10 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Oseltamivir

INTERVENTIONS:
Drug: Baloxavir Marboxil — Given PO
  Other Names: BXM; Xofluza
  Arms: Arm I (oseltamivir, baloxavir marboxil)
Drug: Oseltamivir — Given PO

SUMMARY:
This phase II trial studies the effect of baloxavir in combination with oseltamivir in treating severe influenza infection in patients who have previously received a hematopoietic (blood) stem cell transplant or have a hematological malignancy. Baloxavir is an antiviral drug that inhibits the growth of influenza virus, reduces viral load and prevents further influenza infection. Osetamivir is an antiviral drug that blocks enzymes on the surfaces of influenza viruses, interfering with cell release of complete viral particles. Giving baloxavir in combination with oseltamivir may shorten or decrease the intensity of influenza infection compared to oseltamivir alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To compare the efficacy of baloxavir marboxil (baloxavir) in combination with oseltamivir to oseltamivir monotherapy as measured by changes in influenza viral loads at day 1 from baseline for treatment of severe influenza infections in immunocompromised hosts (such as hematopoietic cell transplant [HCT] recipients and hematological malignancy [HM] patients) and compare the main clinical outcome, complicated hospital stay between the intervention arm and control arm.

SECONDARY OBJECTIVES:

I. To compare the efficacy of baloxavir in combination with oseltamivir to oseltamivir monotherapy as measured by changes in influenza viral loads at day 3, 7, 14 and 30 from baseline.

II. To measure the incidence of baloxavir and oseltamivir resistance, development of lower respiratory tract infections (LRTI), oxygen requirement, respiratory failure, changes in microbiome of the upper airway, length of hospital stay and all-cause mortality at day 30 while on baloxavir and/or oseltamivir in these immunocompromised hosts.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive oseltamivir orally (PO) twice daily (BID) for up to 10 days and baloxavir marboxil PO every 72 hours for a total of 3 doses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive oseltamivir PO BID for up to 10 days in the absence of disease progression or unacceptable toxicity.

After completion of study, patients are followed up at 30 days.

ELIGIBILITY:
Inclusion criteria:

1. Hematopoeitic cell transplant recipients OR hematological malignancy patients
2. Diagnosed with influenza ⱡ
3. Evidence of LRTI* or high risk upper respiratory tract infection (URTI)**

ⱡ A positive multiplex PCR for influenza is required to confirm a diagnosis of influenza infection.

* LRTI will be defined as influenza cases that have evidence of disease below the level of the trachea on either imaging only (possible LRTI), imaging and microbiological evidence of lower airway disease with a bronchoscopy (probable LRTD) or pathological evidence of disease via biopsy (proven LRTI).

** High risk URI will be defined as those cases of influenza that do not have microbiological nor radiological evidence of LRTI, yet they have an immunodeficiency scoring index (ISI) of 3 or greater as defined by Shah D et al (19) for HCT recipients or severe neutropenia (ANC ≤500 cells/ml) and/or lymphopenia (ALC ≤200 cells/ml) for HM patients.

Exclusion criteria:

1. Patient requires mechanical ventilation at time of enrollment
2. Patient is younger than the age of 12 years old
3. The patient is unable to tolerate oral therapy
4. The patient is pregnant at screening ( Positive serum β-HCG (beta-human chorionic gonadotropin) test for women of child-bearing potential).
5. The patient is on a prohibited medication. These include Influenza antiviral drugs with the exception of oseltamivir and baloxavir (such as peramivir, laninamivir, zanamivir, rimantadine, umifenovir or amantadine) and herbal therapies.
6. The patient is unable to consent will be excluded

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Changes in viral loads | On day 0, 1, 3, 7, 14, and 30
  Will be measured via repeat nasopharyngeal swabs at each follow up on day 0, 1, 3, 7, 14 and 30 for influenza quantification.
Incidence of complicated hospital stay | Up to 30 days
  Defined as a hospital admission that was either prolonged (greater than 7 days), requiring intensive care unit level of care or death at day 30 as a result of influenza infection.

SECONDARY OUTCOMES:
Rate of resistance to antiviral agents | Up to 30 days
  Will compare variables between the interventional and control groups using Fischer's exact test or Wilcoxon rank sum test when appropriate.
Progression to lower respiratory tract infections | Up to 30 days
  Will compare variables between the interventional and control groups using Fischer's exact test or Wilcoxon rank sum test when appropriate.
Length of hospital stay | Up to 30 days
  Will compare variables between the interventional and control groups using Fischer's exact test or Wilcoxon rank sum test when appropriate.
Oxygen requirement | Up to 30 days
  Will compare variables between the interventional and control groups using Fischer's exact test or Wilcoxon rank sum test when appropriate.
Rate of respiratory failure | Up to 30 days
  Will compare variables between the interventional and control groups using Fischer's exact test or Wilcoxon rank sum test when appropriate.
30-day mortality | At 30 days
  Will compare variables between the interventional and control groups using Fischer's exact test or Wilcoxon rank sum test when appropriate.
Changes in microbiome diversity | On day 0, 1, 3, 7, 14, and 30
  Analysis of alpha and beta diversity of microbiome will be assessed using Agile Toolkit for Incisive Microbial Analyses. Using Shannon index, we will quantify the alpha diversity of the microbiome. Changes in microbiome diversity will be made by comparing alpha diversity at each time point of sample collection (days 0, 1, 3, 7, 14 and 30).

CONTACTS AND LOCATIONS:
Overall Officials: Roy F Chemaly, MD,MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org